CLINICAL TRIAL: NCT04699617
Title: The Feasibility and Efficacy of an Immersive Virtual Reality Software in Parkinson's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Neurológico Sénior (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: CNS2021-01
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A two-arm, randomized, single-blind (blind rater for primary and secondary outcomes), delayed-start feasibility and efficacy trial.
Who Masked: Outcomes Assessor
Masking Description: single-blind (blind rater for primary and secondary outcomes)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Experimental): The active arm will include 3 days a week of training with the Dolphin 2.0 for 12 consecutive weeks. Each session will have the duration of 60 minutes.
  Interventions: Device: Dolphin 2.0
- Delayed-start control arm (Active Comparator): The delayed-start control arm will have six-weeks of physiotherapy specialized for PD (3 times/week, 60 minutes/session) and six-weeks of 3 days a week of training with the Dolphin 2.0, with sessions of 60 minutes.
  Interventions: Device: Dolphin 2.0

INTERVENTIONS:
Device: Dolphin 2.0 — The Dolphin 2.0 is a platform that runs an immersive virtual reality software, based on an oceanic environment, where players control simulated creatures.

SUMMARY:
The Dolphin 2.0 is a platform that runs an immersive virtual reality software, based on an oceanic environment, where players control simulated creatures (dolphin, orca, axolotl). Video games lead to high levels of motivation and arousal, provide immediate feedback and playback, provide explicit reward and implicit success, and titrate difficulty levels. This encourages the practice of exercise, being an important complement to physiotherapy sessions.

The main goal of this study is to evaluate the feasibility, safety and efficacy of an immersive virtual reality software (Dolphin, 2.0) in Parkinson's disease symptomatic control, in a two-arm, randomized, single-blind (blind rater for primary and secondary outcomes), delayed-start feasibility and efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Parkinson's disease according to MDS criteria;
* Hoehn and Yahr stages between I-III (MED ON);
* Ability to perform the Time Up and Go test in normal pace and without assistance, in less than 11,5 seconds in ON state;
* Stable medication for the past 1 month
* Ability to communicate with the investigator, to understand and comply with the requirements of the study;
* Willing and able to provide written informed consent to participate in the study.

Exclusion Criteria:

* History of falls (1 fall in the 3 previous months);
* Psychiatric major co-morbidity (e.g., major depressive disorder as determined by DSM IV criteria);
* A Montreal Cognitive Assessment (MoCA) score < 21;
* Significant visual or visual-perceptual deficits or neuropsychological impairments that may limit participation in the protocol;
* Having any other neurological/orthopaedic disorders likely to affect gait or exercise capacity, e.g., history of stroke;
* Unstable medical condition including cardiovascular instability in the past 6 months
* Interfering activities performed at high level (sports);
* Inability to correctly respond to the assessment protocol according to the clinician's judgment or lack of support from caregiver for this effect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Time reduction in seconds in the Time Up and Go (TUG) test (early intervention effect) | 6-weeks (T1)
  Early intervention effect: superiority of active versus control group with respect to TUG at 6 weeks

SECONDARY OUTCOMES:
Time reduction in seconds in the TUG test (late intervention effect) | 12-weeks (T2) and 16-weeks (T3)
  Late intervention effect: superiority of active group versus control group with respect to TUG result at 12 and 16-weeks
Change in MDS-UPDRS | Baseline, 6-week, 12-week and 16-week
  Difference between groups in MDS-UPDRS
Change in Mini-best test | Baseline, 6-week, 12-week and 16-week
  Difference between groups in Mini-best test
Change in SCOPA-Cog | at baseline and 16-week
  Difference between groups in SCOPA-Cog
Change in PDQ-39 score | at baseline and and 12-week
  Difference between groups in PDQ-39 score
Change in Clinical Global Improvement | Baseline, 6-week, 12-week and 16-week
  Difference between groups in Clinical Global Improvement
Change in Patient Global Impression - Change | Baseline, 6-week, 12-week and 16-week
  Difference between groups in Patient Global Impression - Change
System Usability Scale | after the 1st session of 1st week and the last sessions of 6th and 12th weeks
  Difference between groups in System Usability Scale
Simulator Sickness Questionnaire | after the 1st session of 1st week and the last sessions of 6th and 12th weeks
  Difference between groups in Simulator Sickness Questionnaire
Number of steps/day | Baseline, 6-week, 12-week and 16-week
  Difference between groups in Patients' level of physical activity (number of steps/day, time spent in each level of activity)
Time spent in each level of activity | Baseline, 6-week, 12-week and 16-week
  Difference between groups in Patients' level of physical activity (number of steps/day, time spent in each level of activity)
Change in BMI | Baseline, 6-week, 12-week and 16-week
  Difference between groups in BMI
Change in Schwab and England scale | at baseline and 12-week
  Difference between groups in Schwab and England scale
Patients' satisfaction and perceived exertion | after the 1st session of 1st week and the last sessions of 6th and 12th weeks
  Difference between groups in Patients' satisfaction and perceived exertion (7-points Likert scale)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Ferreira, MD,PhD, Principal Investigator — CNS - Campus Neurológico
Locations (1):
- Campus Neurológico Sénior, Torres Vedras, Portugal

IPD SHARING:
Plan to Share IPD: No
The methodology followed and the results of the study will be shared at the end through publication in a peer-review journal

REFERENCES:
- [Derived] Pimenta Silva D, Bouca-Machado R, Pona-Ferreira F, Lobo T, Cacho R, Anker R, Krakauer JW, Ferreira JJ. Combining immersive exergaming with physiotherapy in a specialized intensive Parkinson's disease rehabilitation program: a randomized controlled trial. J Neuroeng Rehabil. 2025 Jun 11;22(1):131. doi: 10.1186/s12984-025-01640-w. PMID 40500714
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886